CLINICAL TRIAL: NCT03695393
Title: Stigma, Risk Behaviors and Health Care Among HIV-infected Russian People Who Inject Drugs
Acronym: SCRIPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-38069; R00DA041245 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections; Stigmatization; Substance Use
Keywords: Injection drug use; Stigma; HIV
MeSH Terms: conditions — HIV Infections; Stereotyping; Substance-Related Disorders; Social Stigma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention- ACT Therapy (Experimental): Participants randomized to this group will receive three ACT sessions over 1 month
  Interventions: Behavioral: ACT Therapy
- Standard of Care (No Intervention): Participants in the control group will receive standard care as normally provided to patients by civil society organizations.

INTERVENTIONS:
Behavioral: ACT Therapy — The ACT intervention will consist of three 2-hour group sessions of culturally adapted ACT (intervention) to reduce stigma and related manifestations.Participants are recruited from a civil society organization and all other study procedures take place at a rehabilitation center. The ACT sessions will be scheduled to take place at the rehabilitation center following randomization.The First St. Petersburg Pavlov State Medical University is an alternative location where sessions can be conducted. Sessions will be planned to occur in weekly succession, with a goal of 3 sessions within the first month of study participation.
  Arms: Intervention- ACT Therapy

SUMMARY:
This study is a randomized controlled trial (RCT) among 100 HIV-positive people with injection drug use, which aims to test the feasibility of the SCRIPT intervention and evaluate its effectiveness on the reduction of internalized stigma, as well as entry into substance use treatment or initiation of antiretroviral therapy.

DETAILED DESCRIPTION:
People who inject drugs often experience multiple layers of stigma when they are living with HIV. Stigma is defined as the social exclusion and dehumanization of individuals in an undesirable social category. Interventions to help affected people who inject drugs living with HIV cope with the dual stigma related to HIV and substance use have not been studied specifically in this population. Among people living with HIV, stigma adversely impacts all aspects of the care cascade: timely HIV testing, diagnosis, treatment, adherence and retention in care. Among people who inject drugs, drug use may add to adverse social factors and create particular stigma vulnerability. Russia is a country where people who inject drugs and other HIV key populations are highly stigmatized and face discrimination. Further qualitative findings suggest that in the absence of public anti-stigma campaigns in Russia, stigma reduction interventions should address internalized stigma and their determinants to help affected people cope with the dual stigma. Stigma interventions should be adapted to address not only affected people's shame and guilt, but also their felt hopelessness. These emotions and related feelings such as avoidance and fear of being rejected may negatively affect people's agency and mental health. We are proposing Acceptance and Commitment Therapy (ACT) as a potential behavioral intervention to target the emotions underlying internalized stigma and thus empower affected people. ACT has been shown to increase engagement in addiction care. Its use and efficacy to reduce stigma has not yet been explored among HIV-positive people who inject drugs. The objective of this study, "Stigma, Risk Behaviors and Health Care among HIV-positive Russian People Who Inject Drugs (SCRIPT),"is to implement and evaluate, the feasibility of ACT as an intervention to reduce dual HIV and substance use stigma via a two-armed randomized controlled trial among 100 HIV-positive people who inject drugs. The central hypothesis is that SCRIPT is feasible and can be delivered to decrease HIV and substance use stigma scores.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HIV-positive
* Current injection drug use (past 30 days)
* Not currently on antiretroviral therapy (ART)
* Provision of contact information for two contacts to assist with follow-up
* Address within 100 kilometers of St. Petersburg
* Possession of a telephone (home or cell)
* Able and willing to comply with all study protocols and procedures over 6 months
* Available at the specific days of the week and times that the group sessions will be occurring for the subsequent 3-4 weeks (to ensure that participants randomized into the intervention arm will be able to receive the intervention)

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment resulting in ability to provide informed consent based on research assessor (RA) assessment
* Acute severe psychiatric illness (i.e., answered yes to any of the following: past three month active hallucinations; mental health symptoms prompting a visit to the Emergency Department (ED) or hospital; mental health medication changes due to worsening symptoms; presence of suicidal plans) and research assessor clinical observation (i.e. clinical observation or prior knowledge of severe personality disorder; past three months active mania; past three months active psychosis)
* Enrolled in another research study
* Participated in the pilot portion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Lunze, MD, Principal Investigator — Boston Medical Center
Locations (1):
- First St. Petersburg Pavlov State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luoma JB, Rossi SL, Sereda Y, Pavlov N, Toussova O, Vetrova M, Bendiks S, Kiriazova T, Krupitsky E, Lioznov D, Blokhina E, Lodi S, Lunze K. An acceptance-based, intersectional stigma coping intervention for people with HIV who inject drugs-a randomized clinical trial. Lancet Reg Health Eur. 2023 Mar 20;28:100611. doi: 10.1016/j.lanepe.2023.100611. eCollection 2023 May. PMID 37180745

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention- Acceptance and Commitment Therapy (ACT): Participants randomized to this group will receive three ACT sessions over 1 month
  Acceptance and Commitment Therapy (ACT): The ACT intervention will consist of three 2-hour group sessions of culturally adapted ACT (intervention) to reduce stigma and related manifestations.Participants are recruited from a civil society organization and all other study procedures take place at a rehabilitation center. The ACT sessions will be scheduled to take place at the rehabilitation center following randomization.The First St. Petersburg Pavlov State Medical University is an alternative location where sessions can be conducted. Sessions will be planned to occur in weekly succession, with a goal of 3 sessions within the first month of study participation.
Period: Overall Study
Arm/Group | Intervention- Acceptance and Commitment Therapy (ACT) | Standard of Care
Started | 67 | 33
1-month | 66 | 32
6-month | 64 | 31
Completed | 64 | 31
Not Completed | 3 | 2
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention- ACT Therapy | Standard of Care | Total
Number analyzed (Participants) | 67 | 33 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 33 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.28 (4.87) | 37.67 (6.39) | 38.08 (5.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 16 | 49
  Male | 34 | 17 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  White | 65 | 31 | 96
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 67 | 33 | 100
Education [Count of Participants; unit: Participants]
  Middle school or less | 17 | 10 | 27
  High school/college | 47 | 23 | 70
  Higher education | 3 | 0 | 3
Marital status [Count of Participants; unit: Participants]
  Married/domestic partnership | 43 | 24 | 67
  Long-term relationship but not living together | 4 | 2 | 6
  Single/Divorced/Widowed/Separated | 20 | 7 | 27
HIV internalized stigma [Mean (Standard Deviation); unit: Units on a scale] — Mean HIV internalized stigma score at baseline. Measured via a modified HIV internalized stigma scale, a 7-item questionnaire. Each item had yes/no options. Scores ranged from 0 to 7. Higher scores correspond to higher HIV stigma.
  Units on a scale | 3.31 (1.78) | 3.52 (1.60) | 3.38 (1.72)
Substance use stigma [Mean (Standard Deviation); unit: Units on a scale] — Substance use stigma score between at baseline. Measured via Modified Substance Abuse Self-Stigma Scale, an 12-item questionnaire. Each item was assessed on a 5-point Likert scale. Scores ranged from 12 to 60. Higher scores correspond to higher substance use stigma.
  Units on a scale | 31.40 (7.27) | 32.45 (7.35) | 31.75 (7.28)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Satisfied With the Intervention
Description: Number of participants with satisfaction score of ≥ 3 out of 5. Score determined by an average of a 3-item Likert scale (1-5) questionnaire, developed by the study team.
Time Frame: 1 month
Population: Participants who completed the 1-month assessment and attended at least one session. 64 of the 66 intervention participants completed the 1-month assessment AND at least one intervention session.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 64 | 0
Participants | 61 | 0

2. Primary Outcome: Change in HIV Stigma Score
Description: Mean change in HIV internalized stigma score between baseline and 1 month. Measured via a modified HIV internalized stigma scale, a 7-item questionnaire. Each item had yes/no options. Scores ranged from 0 to 7. Higher scores correspond to higher HIV stigma.
Time Frame: baseline, 1 month
Population: Participants who completed the 1-month assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 66 | 32
units on a scale | 0.45 (1.42) | -0.06 (1.05)

3. Primary Outcome: Change in Substance Use Stigma
Description: Mean change in substance use stigma score between baseline and 1 month. Measured via Modified Substance Abuse Self-Stigma Scale, an 12-item questionnaire. Each item was assessed on a 5-point Likert scale. Scores ranged from 12 to 60. Higher scores correspond to higher substance use stigma.
Time Frame: baseline, 1 Month
Population: Participants who completed the 1-month assessment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 66 | 32
Units on a scale | -1.42 (7.14) | 0.06 (7.81)

4. Secondary Outcome: Number of Participants Who Participated in the Intervention
Description: Defined as the number of participants who participated in three ACT intervention sessions
Time Frame: Throughout the study to completion at 6 months
Population: Only intervention arm participants analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 67 | 0
Participants | 54 | 0

5. Secondary Outcome: Overall Fidelity to Intervention
Description: Defined using the Adherence Raters' Manual for Stigma Treatment Study to rate the recorded intervention tapes. This outcome reports the number of intervention segments that meet adequate fidelity. Overall fidelity rated on a score of 1 (low) to 5 (high). Score of a 3 or above was considered adequate fidelity.
Time Frame: Throughout the study to completion at 6 months
Population: Each intervention session was divided into 3 segments, totaling to 9 segments over 3 sessions. The first segment was discarded, as it only included introductions and no intervention content. The total number of segments throughout the intervention was 104 (8 segments of 13 groups). 30% of these segments were randomly selected to code to assess for fidelity, which resulted in 33 segments coded. This outcome is assessing the intervention segments, not the participants.
Measure: Count of Units; unit: Intervention segments
Units Other Than Participants: Intervention segments
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 67 | 0
Number analyzed (Intervention segments) | 33 | 0
Intervention segments | 33 | 0

6. Secondary Outcome: Initiation of HIV Care
Description: Defined as self-report of antiretroviral therapy (ART) initiation in the past 6 months.
Time Frame: 6 months
Population: Participants who completed the 6-month assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 64 | 31
Participants | 13 | 1

7. Secondary Outcome: Engagement in Substance Use Care
Description: Defined as self-report of treatment of a substance use disorder in an outpatient clinic, inpatient setting, or attendance of 12-step recovery program in the past 6 months.
Time Frame: 6 months
Population: Participants who completed the 6-month assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 64 | 31
Participants | 15 | 2

8. Secondary Outcome: Change in the Total Number of Injections in the Previous 30 Days
Description: Defined as self-report of any change in injection drug use in the previous 30 days measured via a modified Risk Behavior Survey. Participants report total number of injections in the past 30 days.
Time Frame: baseline, 6 months
Population: Participants who completed the 6-month assessment
Measure: Mean (Standard Deviation); unit: Number of injections
Arm/Group | Intervention- ACT Therapy | Standard of Care
Number analyzed (Participants) | 64 | 31
Number of injections | -1.78 (14.60) | 7.16 (22.34)

9. Other Pre Specified Outcome: Depression
Description: Measured via the Patient Health Questionnaire-9, a 9-item questionnaire with higher scores corresponding to greater depression severity.
Time Frame: 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Anxiety
Description: Measured via the Generalized Anxiety Disorder-7 scale, a 7-item questionnaire with higher scores corresponding to greater anxiety severity.
Time Frame: 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Intersectional Stigma
Description: Measured by both substance use stigma and HIV stigma scales, with high scores on both indicating intersectional stigma
Time Frame: 6 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Psychological Flexibility
Description: Measured via Acceptance and Action Questionnaire - Substance Abuse, an 18-item questionnaire. Higher scores correspond to higher psychological flexibility
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the 6-month study period.
Arm/Group | Intervention- ACT Therapy | Standard of Care
All-Cause Mortality (participants affected / at risk) | 3/67 | 1/33
Serious Adverse Events (participants affected / at risk) | 5/67 | 1/33
Other Adverse Events (participants affected / at risk) | 2/67 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention- ACT Therapy (N=67) | Standard of Care (N=33)
Hospitalization due to HIV progression (Immune system disorders) | 1 (1) | 0 (0)
Hospitalization due to pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Death due to stroke (Nervous system disorders) | 0 (0) | 1 (1)
Death due to cerebral edema (Nervous system disorders) | 2 (2) | 0 (0)
Death due to cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention- ACT Therapy (N=67) | Standard of Care (N=33)
HIV progression (Immune system disorders) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03695393/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT03695393/ICF_001.pdf